CLINICAL TRIAL: NCT04897308
Title: Shoulder Adhesive Capsulitis ; Comparison Between Three Theraputic Approaches
Brief Title: Best Treatment Modality of Frozen Shoulder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Shorouk Ayman Mohamed, Resident doctor, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Soh-Med-21-05-04
Record Dates: First submitted 2021-05-16; First posted 2021-05-21 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Shoulder Adhesive Capsulitis
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Suprascapular nerve block (Active Comparator): This group will include will under go suprascapularnerve block as following :10 ml of .5% bupivacaine and 2 ml of methylpradnisolon 40mg/ml
  Interventions: Procedure: Local injection of shoulder joint
- Hydrodilatation of shoulder capsule (Active Comparator): This group will undergo intraarticular hydrodilatation by injection of :first lidocaine10ml%followed by 1ml of methylprednisolon 40mg/ml and finally 20ml of .9 % sodium chloride slowly in the gleno humeral joint
  Interventions: Procedure: Local injection of shoulder joint
- Hydrodilatation of shoulder interval (Active Comparator): This group will undergo interval hydrodilatation by injection of :first mepivacaine 10ml folowed by 20ml of sterile water slowly in the shoulder interval
  Interventions: Procedure: Local injection of shoulder joint

INTERVENTIONS:
Procedure: Local injection of shoulder joint — Under ultrasound guidance , local shoulder joint injection will be done

SUMMARY:
This study will compare between the effect of three treatment modalities of shoulder adhesive capsulitis to hilight the best technique to improve pain and range of motion outcome measures .

ELIGIBILITY:
Inclusion Criteria:

* gross limitation of passive shoulder movement
* pain interfering with daily activities
* painful restiction of active and passive movement of shoulder

Exclusion Criteria:

* presence of degenerative pathology
* fracture
* contraindication to steroid injection
* deformity affecting upper limb
* history of previous shoulder injection in the past 4 weeks

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Improvement in range of motion of shoulder joint | 12 weeks efter intervention
  Improvement will be measured by measuring active and passive range of motion
Improvement in pain | 12 weeks after intervention
  Improvement will be measured by VAS ( visual auditory assessment )

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag faculty, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No